CLINICAL TRIAL: NCT05132218
Title: Prospective Exploratory Real World Study of Ensatinib in alK-positive Patients Undergoing Initial Treatment for Advanced Non-small Cell Lung Cancer
Brief Title: Ensatinib in alK-positive Patients Undergoing Initial Treatment for Advanced Non-small Cell Lung Cancer
Acronym: EFLRWR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jun Zhao, Professor, Peking University Cancer Hospital & Institute
Other Study IDs: BD-EN-IV002
Record Dates: First submitted 2021-10-26; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: ALK Positive; NSCLC Stage IIIB; NSCLC Stage IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. The patient's tumor tissue sample before taking Ensatinib
  2. The patient's baseline blood sample within the first week before taking Ensantinib
  3. Blood samples of patients 4-6 weeks after taking Ensatinib
  4. Blood samples within 4 weeks after the patient's disease progression
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ensatinib for treated patients with ALK-positive advanced non-small cell lung cancer: Ensatinib 225mg QD Until the disease progresses or intolerance
  Interventions: Drug: Ensatinib

INTERVENTIONS:
Drug: Ensatinib — Prospective, exploratory, single-arm, multi-center, real-world research
  Other Names: BD-EN-IV002

SUMMARY:
The experimental design is exploratory, single-arm, multi-center, real-world research.

Ensatinib 225mg qd A prospective and exploratory real-world study of Ensatinib for ALK-positive advanced non-small cell lung cancer patients Test purposes Exploring the real world, Ensatinib is effective for the newly treated ALK+ advanced NSCLC

1. Efficacy and safety;
2. The relationship between molecular mechanism and curative effect;
3. Ensatinib resistance mechanism;

DETAILED DESCRIPTION:
Enrolled patients:

1. stage IIIB or stage IV NSCLC
2. Each center confirmed ALK+ by tissue samples (Abbott FISH, VENTANA ALK D5F3, NGS method confirmation);
3. Without any ALK-TKI treatment; Study endpoint

Primary endpoint:

According to the RECIST1.1 standard, the progression-free survival (PFS) assessed by the investigator;

Secondary endpoint:

According to the RECIST1.1 standard, the objective response rate (ORR) evaluated by the investigator; the time to treatment failure (TTF); according to the RECIST1.1 standard, the ORR and PFS of patients with different ALK fusion subtypes evaluated by the investigator; total Lifetime (OS); safety;

Exploratory endpoint:

The correlation between the biomarkers in blood or/and tissue samples and the efficacy of Ensatinib; the resistance mechanism of Ensatinib;

The sample size is determined:

The plan is to analyze 60-80 patients with EML4-ALK fusion v1 and v3 subtypes. Based on the proportion of patients with both subtypes in ALK-positive patients, the proportion is about 40%. Based on the 20% dropout rate, the plan is to include ALK without distinction. 180 patients with fusion subtype; statistical methods:

ELIGIBILITY:
Inclusion Criteria:

1. stage IIIB or stage IV NSCLC by histology or cytology;
2. All centers confirmed ALK positive by tissue samples (Abbott FISH, VENTANA ALK D5F3, NGS method confirmation);
3. Without any ALK-TKI treatment;
4. Voluntarily and capable of following the trial and follow-up procedures;
5. Able to understand the nature of the trial, and be able to complete the signing of a written informed consent form.

Exclusion Criteria:

* 1. Pereceived any ALK-TKI treatment ; 2. Received any chemotherapy within 4 weeks, or underwent major surgery or radiotherapy within the last 14 days; 3. The investigator believes that the patient is not suitable for Ensatinib treatment.

Had a stem cell or organ transplant. 4. Having serious cardiovascular disease, including but not limited to: 5.Sino - QTcF interval ≥450 ms or other significant ECG abnormalities. According to the study, researchers either ruled that hypertension was poorly controlled (systolic blood pressure >160 mmHg or diastolic blood pressure >100mmHg).

6. Dysphagia, active gastrointestinal disease, or other disease that significantly affects drug absorption, distribution, metabolism, and excretion.

7. Previous history of interstitial lung disease, drug-induced interstitial lung disease, radioactive pneumonia requiring steroid treatment, or any indication of clinically active interstitial lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Single arm real world study of non-small cell lung cancer; stage IIIB or stage IV ALK positive NSCLC；
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2021-10-19 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 2021.09.27-2024.12.30

SECONDARY OUTCOMES:
overall survival | 2021.09.27-2024.12.30
Time-to-TreatmentFailure | 2021.09.27-2024.12.30

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China